CLINICAL TRIAL: NCT00127231
Title: Brief Alcohol Intervention in HIV+ Women
Brief Title: Brief Therapy Intervention for Heavy/Hazardous Drinking in HIV-Positive Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAAMCC014500; R01AA014500 (NIH); K23AA015313 (NIH)
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: HIV Infections; Alcoholism
Keywords: Controlled Clinical Trials, Randomized; Alcohol Consumption; Behavioral Research; HIV; Alcohol Abuse
MeSH Terms: conditions — HIV Infections; Alcoholism; Alcohol Drinking | interventions — Ethanol; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Brief Intervention (Experimental): The brief intervention will include two sessions that review drinking patterns and behavior change strategies as well as two telephone calls to reinforce session content.
  Interventions: Behavioral: Brief alcohol intervention based on Project Treat
- 2 Standard Care Arm (Active Comparator)
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Brief alcohol intervention based on Project Treat — The brief intervention will include two sessions that review drinking patterns and behavior change strategies as well as two telephone calls to reinforce session content.
  Arms: 1 Brief Intervention
Behavioral: Standard care — Hazardous/binge female drinkers will be identified in the Johns Hopkins Hospital HIV clinic and will be randomized to brief intervention or standard care. Outcome measures will include: alcohol/drug use, engagement in an on-site alcohol support group and other substance abuse treatment services, HIV-risk behaviors, HIV disease markers and treatment compliance, and psychiatric symptoms.
  Arms: 2 Standard Care Arm

SUMMARY:
The purpose of this study is to determine whether two brief counseling sessions reduce drinking and improve health outcomes in HIV-positive women who drink at heavy/hazardous levels. Also, the study seeks to compare hazardous drinking versus nonhazardous drinking women on a variety of alcohol, HIV and life quality outcome measures.

DETAILED DESCRIPTION:
Heavy alcohol use negatively impacts HIV/AIDS in several important ways. It increases HIV-risk behaviors, impairs the immune system and accelerates HIV disease progression. Heavy alcohol use also interferes with HIV care compliance, including appointment attendance and medication adherence.

Women are particularly important targets for alcohol use interventions. The threshold for harmful alcohol effects is strikingly low in women, with two drinks per day placing women at risk for negative health consequences. Heavy/hazardous alcohol use is less likely to be detected in women receiving health services. Women may be less likely to seek and or engage in alcohol treatment services, making nontraditional care settings particularly important for reaching this population.

This proposal tests the utility of a brief alcohol intervention for HIV+ women delivered in a medical setting. Hazardous/binge female drinkers will be identified in the Johns Hopkins Hospital HIV clinic and will be randomized to brief intervention or standard care. The brief intervention will include two sessions that review drinking patterns and behavior change strategies as well as two telephone calls to reinforce session content. In addition, a comparison group of nonhazardous drinking, HIV+ women will be recruited. Outcome measures will include: alcohol/drug use, engagement in an on-site alcohol support group and other substance abuse treatment services, HIV-risk behaviors, HIV disease markers and treatment compliance, and psychiatric symptoms.

The investigators hypothesize that women who receive the brief intervention will report lower mean weekly alcohol consumption and fewer heavy drinking episodes than women in standard care. The investigators also predict that women who receive brief intervention will adhere to their HIV medications and keep their health care appointments more consistently, and have improved HIV-related health outcomes. Finally, the investigators hypothesize that nonhazardous drinkers will have fewer psychiatric symptoms and better quality of life than hazardous drinking women.

Comparison(s): Standard HIV care

ELIGIBILITY:
Inclusion Criteria:

* Heavy/hazardous drinking levels (i.e., consuming 8 or more drinks per week, or have reported at least two heavy drinking occasions [4 or more drinks/drinking episode] in the last six months, or score positively on the CAGE or T-ACE).
* HIV-positive
* Receiving HIV care in Johns Hopkins Hospital (JHH) Moore Clinic

Exclusion Criteria:

* Actively psychotic and other severe mental health symptoms
* Current enrollment in alcohol or drug treatment
* Current enrollment in Hopkins psychiatric services
* Pregnancy (because of the ethical concern of randomization to standard care)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2007-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. McCaul, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 Brief Intervention | 2 Standard Care Arm
Started | 74 | 74
Completed | 68 | 68
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Brief Intervention | 2 Standard Care Arm | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at baseline assessment (Years)
  years | 46.27 (7.07) | 44.86 (9.1) | 45.56 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex at baseline assessment
  Participants
    Female | 74 | 74 | 148
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race at baseline assessment
  Participants
    American Indian or Alaska Native | 0 | 2 | 2
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 67 | 60 | 127
    White | 7 | 12 | 19
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 74 | 74 | 148
Employment % [Count of Participants; unit: Participants] — Current employment status at baseline assessment
  Participants
    Working part-time or full-time | 21 | 28 | 49
    Unemployed | 53 | 46 | 99
Income, Continuous [Mean (Standard Deviation); unit: dollars] — Annual income at baseline assessment (US dollars)
  dollars | 8497.38 (7166.03) | 8189.19 (7239.17) | 8343.28 (7202.60)
Undetectable HIV-1 RNA % [Count of Participants; unit: Participants]
  Undetectable HIV-1 RNA (<50 copies) | 29 | 31 | 60
  Detectable HIV-1 RNA | 45 | 43 | 88
CD4 count, Continuous [Mean (Standard Deviation); unit: cells/mm3] | 398.11 (269.02) | 393.24 (236.78) | 395.68 (252.9)
AUDIT score, continuous [Mean (Standard Deviation); unit: units on a scale] — Score on the Alcohol Use Disorders Identification Test (AUDIT) at baseline assessment. The AUDIT ranges from 0 (minimum) to 40 (maximum). The higher the score, the more likely it is that the individual has an alcohol use disorder.
  units on a scale | 11.9 (8.7) | 12.3 (8.9) | 12.1 (8.8)
Total number of drinking days out of the past 90 days [Mean (Standard Deviation); unit: days] | 34.03 (29.47) | 30.45 (27.57) | 32.24 (28.52)
Number of standard drinks per episode, continuous [Mean (Standard Deviation); unit: standard drinks] — A standard drink is any drink that contains about 14 grams of pure alcohol. One standard drink is typically considered to be 12 fluid ounces of beer, 4 - 5 fluid ounces of wine, or 1.5 fluid ounces of 80 proof liquor.
  standard drinks | 9.69 (9.13) | 9.55 (6.42) | 9.62 (7.78)
Number of participants with illicit drug use in past 6 months [Count of Participants; unit: Participants] | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinking Days Out of the Past 90 Days
Time Frame: Baseline through 1 year follow-up
Population: All randomized participants were included in analyses although 6 participants from each arm did not complete the study due to loss to follow up
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 1 Brief Intervention | 2 Standard Care Arm
Number analyzed (Participants) | 74 | 74
days
  Baseline | 34.03 (29.47) | 30.45 (27.57)
  3-month follow-up: number analyzed (Participants) | 55 | 57
  3-month follow-up | 13.58 (19.89) | 20.22 (25.27)
  6-month follow-up: number analyzed (Participants) | 62 | 62
  6-month follow-up | 14.42 (22.20) | 24.48 (26.78)
  12-month follow-up: number analyzed (Participants) | 64 | 64
  12-month follow-up | 15.96 (24.07) | 20.83 (27.53)
Statistical Analysis 1: Comparison: 1 Brief Intervention vs 2 Standard Care Arm; Drinking frequency was analyzed using a generalized binomial mixed-effects model with the logit link function and a random intercept. The use of a binomial distribution was indicated for this analysis because the outcome was assessed using a 90-day TLFB interview, which has a cap at 90 days; Test type: Equivalence; p < 0.005, Mixed Models Analysis; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.23 to 0.75]

2. Primary Outcome: Number of Binge Drinking Days Out of the Past 90 Days
Description: Number of days during the past 90 days on which women drank more than 3 standard drinks
Time Frame: Baseline through 12 month follow-up
Population: Not all subjects participated in every follow-up interview.
Measure: Mean (Standard Deviation); unit: days out of past 90 days
Arm/Group | 1 Brief Intervention | 2 Standard Care Arm
Number analyzed (Participants) | 74 | 74
days out of past 90 days
  Baseline | 24.91 (26.99) | 26.71 (28.55)
  3-month follow-up: number analyzed (Participants) | 55 | 57
  3-month follow-up | 7.68 (13.75) | 13.95 (22.11)
  6-month follow-up: number analyzed (Participants) | 62 | 62
  6-month follow-up | 12.07 (21.61) | 16.14 (23.63)
  12 month follow-up: number analyzed (Participants) | 64 | 64
  12 month follow-up | 12.76 (23.42) | 13.23 (20.40)

3. Secondary Outcome: HIV Clinic Appointment Adherence (Kept/Scheduled Appointments)
Description: the % of kept appointments out of scheduled appointments was determined for each participant, and then averaged for the set of participants at each time point
Time Frame: baseline through 1 year follow-up
Measure: Mean (Standard Deviation); unit: percentage of kept/scheduled appointment
Arm/Group | 1 Brief Intervention | 2 Standard Care Arm
Number analyzed (Participants) | 74 | 74
percentage of kept/scheduled appointment
  Baseline | 63.40 (23.47) | 58.59 (23.66)
  3-month follow-up | 70.11 (25.15) | 60.57 (33.69)
  6-month follow-up | 67.87 (28.57) | 62.22 (33.98)
  12-month follow-up | 63.33 (23.82) | 56.63 (27.91)

4. Secondary Outcome: % of Patients Currently on Antiretroviral Therapy
Description: number of participants who are currently receiving antiretroviral therapy/total number of participants
Time Frame: baseline through 1 year follow-up
Measure: Number; unit: percentage of participants
Arm/Group | 1 Brief Intervention | 2 Standard Care Arm
Number analyzed (Participants) | 74 | 74
percentage of participants
  Baseline | 72.97 | 67.57
  3-month follow-up | 78.18 | 68.42
  6-month follow-up | 75.81 | 70.97
  12-month follow-up | 84.38 | 76.56

5. Secondary Outcome: Number of Days in Past 90 Days on Which Participants Reported Having Unprotected Vaginal Sex
Description: Number of days in the past 90 days on which participants reported having unprotected vaginal sex
Time Frame: Baseline to 12 month follow-up
Population: Not all subjects participated in every follow-up interview.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 1 Brief Intervention | 2 Standard Care Arm
Number analyzed (Participants) | 74 | 74
days
  Baseline | 2.68 (8.61) | 3.31 (9.21)
  3-month follow-up: number analyzed (Participants) | 55 | 57
  3-month follow-up | 2.56 (12.15) | 3.06 (10.31)
  6-month follow-up: number analyzed (Participants) | 62 | 62
  6-month follow-up | 2.31 (7.83) | 1.35 (4.54)
  12-month follow-up: number analyzed (Participants) | 64 | 64
  12-month follow-up | 1.59 (5.11) | 4.74 (13.78)

ADVERSE EVENTS:
Time Frame: Baseline to 12 month follow-up
Arm/Group | 1 Brief Intervention | 2 Standard Care Arm
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No